CLINICAL TRIAL: NCT04715477
Title: Intensive Care Anxiety in SARS-CoV-2 (COVID 19) Patients
Brief Title: Intensive Care Anxiety in SARS-CoV-2 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, İLKE KÜPELİ, assoc. prof., Derince Training and Research Hospital
Other Study IDs: derince TRH 2
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital Anxiety Depression Measure: Hospital Anxiety Depression Measure
  Interventions: Behavioral: Hospital Anxiety Depression Measure

INTERVENTIONS:
Behavioral: Hospital Anxiety Depression Measure — Hospital Anxiety Depression Measure

SUMMARY:
It should be known by the clinician that COVID-19 patients are prone to anxiety, and these disorders need to be properly diagnosed and addressed to improve prognosis, shorten hospital stay and avoid long-term mental health problems.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* COVID PCR +,
* admitted to intensive care,
* conscious, cooperative patients

Exclusion Criteria:

* Having hearing and speaking problems,
* Can't speak Turkish or English,
* who do not have the cognitive level to understand and answer the questions,
* Communication problems such as dementia and Alzheimer's,
* patients receiving sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Co-operative patients over 18 years of age, with COVID PCR + admission to intensive care unit, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-17 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
intensive care Anxiety | 3 month
  Hospital Anxiety Depression scale

CONTACTS AND LOCATIONS:
Overall Officials: ilke kupeli, Principal Investigator — Derince Training and Research Hospital
Locations (1):
- İlke Küpeli, İzmit, Kocaeli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Deng J, Zhou F, Hou W, Silver Z, Wong CY, Chang O, Huang E, Zuo QK. The prevalence of depression, anxiety, and sleep disturbances in COVID-19 patients: a meta-analysis. Ann N Y Acad Sci. 2021 Feb;1486(1):90-111. doi: 10.1111/nyas.14506. Epub 2020 Oct 2. PMID 33009668
- [Result] Rogers JP, Chesney E, Oliver D, Pollak TA, McGuire P, Fusar-Poli P, Zandi MS, Lewis G, David AS. Psychiatric and neuropsychiatric presentations associated with severe coronavirus infections: a systematic review and meta-analysis with comparison to the COVID-19 pandemic. Lancet Psychiatry. 2020 Jul;7(7):611-627. doi: 10.1016/S2215-0366(20)30203-0. Epub 2020 May 18. PMID 32437679
- [Result] 3. Aydemir Ö, Güvenir T, Küey L, Kültür S. Hastane Anksiyete ve Depresyon Ölçeği Türkçe Formunun Geçerlik Güvenilirlik Çalışması. Türk Psikiyatri Dergisi 1997;8:280-287.
- [Derived] Kupeli I, Kara MY, Yakin I, Caglayan AC. Anxiety and depression in the first 24 h in COVID-19 patients who underwent non-invasive mechanical ventilation in the intensive care unit. Ir J Med Sci. 2022 Oct;191(5):2291-2295. doi: 10.1007/s11845-021-02808-8. Epub 2021 Oct 19. PMID 34664224